CLINICAL TRIAL: NCT05191836
Title: Assessing an Active Distracting Technique During Pulpotomy in Primary Mandibular Molar.
Brief Title: Pain and Anxiety Reducing During Dental Treatment in Children Using Video Game on Tablet Device With Joystick.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Pedo-08-2019
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Pulpotomy; Dental Caries; Primary Teeth
Keywords: Children's dental anxiety; video game
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulpotomy in primary mandibular molars by using video game distraction. (Experimental)
  Interventions: Behavioral: Evaluation of the effectiveness of Video Game Distraction in the management of anxious pediatric patients during dental treatment
- Pulpotomy in primary mandibular molars by using audio visual distraction. (Experimental)
  Interventions: Behavioral: Evaluation of the effectiveness of Audio Video Distraction in the management of anxious pediatric patients during dental treatment
- Pulpotomy in primary mandibular molars without using any type of distraction aids (Other)
  Interventions: Other: Evaluation of the anxiety in pediatric patients during dental treatment without using any type of distraction aids

INTERVENTIONS:
Behavioral: Evaluation of the effectiveness of Video Game Distraction in the management of anxious pediatric patients during dental treatment — The child will be provided dental treatment during watching video game.The Behavior Rating Scale "HOUPT" will be measured four times: directly when the patient seated comfortably on the dental chair, after anesthesia, after pulpotomy, and when the treatment completed.
  All child patients will ask to choose a face that describe their status from one of the Simplified Wong Baker faces scale in the same four times.
  Arms: Pulpotomy in primary mandibular molars by using video game distraction.
Behavioral: Evaluation of the effectiveness of Audio Video Distraction in the management of anxious pediatric patients during dental treatment — The child will be provided dental treatment during audio video distraction.The Behavior Rating Scale "HOUPT" will be measured four times: directly when the patient seated comfortably on the dental chair, after anesthesia, after pulpotomy, and when the treatment completed.
  The child will be provided dental treatment during watching video game. All child patients will ask to choose a face that describe their status from one of the Simplified Wong Baker faces scale in the same four times.
  Arms: Pulpotomy in primary mandibular molars by using audio visual distraction.
Other: Evaluation of the anxiety in pediatric patients during dental treatment without using any type of distraction aids — The child will be provided dental treatment without using any type of distraction aids.The Behavior Rating Scale "HOUPT" will be measured four times: directly when the patient seated comfortably on the dental chair, after anesthesia, after pulpotomy, and when the treatment completed.
  The child will be provided dental treatment during watching video game. All child patients will ask to choose a face that describe their status from one of the Simplified Wong Baker faces scale in the same four times.
  Arms: Pulpotomy in primary mandibular molars without using any type of distraction aids

SUMMARY:
The aim of this study is to evaluate the effectiveness of two different distraction techniques (Audio Video Distraction /Video Game Distraction) in the management of anxious pediatric patients during dental treatment.

Group A: pulpotomy in temporary inferior molar will be treated with using video game on tablet device with wireless joystick and wireless headphone

Group B: pulpotomy in temporary inferior molar will be treated with using AV tablet and wireless headphone.

Group C (Control group): pulpotomy in temporary inferior molar will be treated with basic behavior guidance techniques and without using any type of distraction aids.

All of the children who experienced a pulpotomy in temporary inferior molar with/without distraction will be assessed by using a combination of measures: Simplified Wong-Baker faces(self-report), and "HOUPT" Behavior Rating Scale for Movement - Crying - Overall Behavior (nonself-report).

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of two types of distraction aids that contain video game on tablet device with wireless (joystick and headphone) along with audio video distraction using tablet device and wireless headphone.

Pain and anxiety will be evaluated during pulpotomy in temporary inferior molar using two behavioral scales, Simplified Wong-Baker faces (self-report), and "HOUPT" Behavior Rating Scale for Movement - Crying - Overall Behavior (nonself-report).

The Behavior Rating Scale "HOUPT" will be measured four times: directly when the patient seated comfortably on the dental chair, after anesthesia, after pulpotomy, and when the treatment completed.

All child patients will ask to choose a face that describe their status from one of the Simplified Wong Baker faces scale in the same four times.

ELIGIBILITY:
Inclusion Criteria:

1. age between 6 and 10 years.
2. no previous dental experience.
3. definitely positive or positive ratings of Frank scale.
4. Need of pulpotomy in temporary inferior molar.

Exclusion Criteria:

1. previous dental experience
2. systematic or mental disorders.
3. definitely negative or negative ratings of Frankel scale
4. don't need of pulpotomy in temporary inferior molar

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Pain levels | 20 minutes following the end of the treatment session
  Pain levels will be measured by using a self-reported simplified Wong-Baker faces pain scale:
  0 no pain - 1 mild pain - 2 moderate pain - 3 worst pain
Anxiety levels | 20 minutes following the end of the treatment session
  Anxiety levels will be measured by using the "HOUPT" Behavior Rating Scale for Movement - Crying - Overall Behavior:
  For movement: 1 violent movement - 2 continuous movement - 3 controllable movement - 4 no movement.
  For crying: 1 hysterical crying - 2 continuous crying - 3 mild crying - 4 no crying.
  For overall behavior: 1 no treatment - 2 treatment interrupted, only partial treatment completed - 3 treatment interrupted, but eventually all completed - 4 difficult, but all treatment performed - 5 some limited crying or movement - 6 no crying or movement.

CONTACTS AND LOCATIONS:
Overall Officials: Ekram M Al-sibai, DDs, Principal Investigator — MSc student in Pedodontics, University of Damascus; Nada G Bshara, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minute M, Badina L, Cont G, Montico M, Ronfani L, Barbi E, Ventura A. Videogame playing as distraction technique in course of venipuncture. Pediatr Med Chir. 2012 Mar-Apr;34(2):77-83. doi: 10.4081/pmc.2012.64. PMID 22730632
- [Background] Abdelmoniem SA, Mahmoud SA. Comparative evaluation of passive, active, and passive-active distraction techniques on pain perception during local anesthesia administration in children. J Adv Res. 2016 May;7(3):551-6. doi: 10.1016/j.jare.2015.10.001. Epub 2015 Oct 19. PMID 27222759
- [Background] Attar RH, Baghdadi ZD. Comparative efficacy of active and passive distraction during restorative treatment in children using an iPad versus audiovisual eyeglasses: a randomised controlled trial. Eur Arch Paediatr Dent. 2015 Feb;16(1):1-8. doi: 10.1007/s40368-014-0136-x. Epub 2014 Nov 22. PMID 25416522
- [Background] Patel A, Schieble T, Davidson M, Tran MC, Schoenberg C, Delphin E, Bennett H. Distraction with a hand-held video game reduces pediatric preoperative anxiety. Paediatr Anaesth. 2006 Oct;16(10):1019-27. doi: 10.1111/j.1460-9592.2006.01914.x. PMID 16972829
- [Background] Millett CR, Gooding LF. Comparing Active and Passive Distraction-Based Music Therapy Interventions on Preoperative Anxiety in Pediatric Patients and Their Caregivers. J Music Ther. 2018 Jan 13;54(4):460-478. doi: 10.1093/jmt/thx014. PMID 29253180
- [Background] Arikan A, Esenay FI. Active and Passive Distraction Interventions in a Pediatric Emergency Department to Reduce the Pain and Anxiety During Venous Blood Sampling: A Randomized Clinical Trial. J Emerg Nurs. 2020 Nov;46(6):779-790. doi: 10.1016/j.jen.2020.05.004. Epub 2020 Jul 22. PMID 32711948